CLINICAL TRIAL: NCT01161888
Title: Effect of Topical Imiquimod on Lentigo Maligna
Acronym: LIMIT-1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jerry Marsden (Other)
Collaborators: Department of Health, United Kingdom (Other Government)
Responsible Party: Sponsor-Investigator, Jerry Marsden, Consultant Dermatologist, University Hospital Birmingham NHS Foundation Trust
Organization: University Hospital Birmingham NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIMIT-1
Record Dates: First submitted 2010-06-24; First posted 2010-07-14 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2010-05

CONDITIONS: Lentigo Maligna
MeSH Terms: conditions — Hutchinson's Melanotic Freckle | interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Imiquimod — 250mg sachets to be applied at a start dose of 5 days a week. Dose will be adjusted using an algorithm according to tolerability.
  Other Names: Aldara 5% cream

SUMMARY:
The purpose of this study is to determine if topical imiquimod is effective in the pathological complete regression of lentigo maligna.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of lentigo maligna (LM) (acquired pigmented macule present for more than 12 months with no change in skin surface texture or contour, no palpability, diameter >10 mm, sited on the head or neck). The lower anatomical limit is the root of the neck - a line joining the medial end of the clavicles with the medial insertion of trapezius.
* Histological findings consistent with LM (increased numbers of atypical melanocytes confined to the epidermis, sun damaged skin) in one or more 4mm punch biopsies(s) from the darkest area, reported by a pathologist with expertise in the diagnosis of melanocytic lesions, and part of a recognised NHS skin cancer Multi-Disciplinary Team.
* The upper limit of the lesion is not defined by size, but it must be suitable for complete surgical excision using a 5 mm lateral margin.
* The outline of the lesion must be easily defined visually in daylight around its entire circumference.
* Patient fit enough and willing to undergo surgery as required by the protocol.

Exclusion Criteria:

* Clinical or histological evidence of invasive melanoma including any palpability of the lesion, or clinical and/or histological evidence of regression or dermal invasion
* Aged less than 45 years
* Recurrent LM - the index lesion must not have been previously treated
* Life expectancy of less than 12 months
* Other skin lesions which may compromise the ability to complete this study, such as co-existing or adjacent melanoma or non-melanoma skin cancer. Co-existing adjacent actinic keratoses would not exclude the patient from the study
* Women of childbearing potential, who are pregnant, plan to become pregnant during their study participation or breastfeeding.
* Unable to give informed consent.
* Hypersensitivity to imiquimod or to any of the excipients (methylhydroxybenzoate (E218), propylhydroxybenzoate (E216), cetyl alcohol and stearyl alcohol).
* Taking immunosuppressive medication.
* Taking part in any other intervention study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Pathological complete regression (PCR) in the mapped biopsied and resected LM using 2 mm slices. | Results available at 1-2 week post surgery follow up visit.

SECONDARY OUTCOMES:
Clinical assessment of response after imiquimod treatment | Assessed at 12 week treatment visit and 1-2 week post surgery follow up
  The pathological response in the entire resected lesion will be compared with that predicted from clinical examination and biopsies taken before surgery, post imiquimod treatment. We will assess whether adequate surgical margins can be determined using clinical maps. It is essential to know the accuracy of the method of clinical assessment of response.
Clinical feasibility of imiquimod treatment | Tolerability will be assessed during treatment period of 12 weeks
  Number of reported local adverse reactions and systemic adverse reactions; adherence to treatment schedule and acceptability of imiquimod treatment.
Number of consultations with NHS staff during imiquimod treatment | Assessed up to week 12 visit
Frequency of functional T cell responses recognising peptide epitopes in melanocyte differentiation and cancer-testis antigens. | Assessed with baseline and 12 week visit samples.
  Circulating immune responses to proteins expressed within melanoma will be measured using blood draws taken before imiquimod treatment and after completion of imiquimod therapy but before surgery. The demonstration of a circulating immune response would be an important finding that would strongly support the investigation of imiquimod as primary therapy for melanoma, even if coupled with subsequent surgery because of the potential for such an immune response to be preventative against recurrence or invasive disease.
Measurement of hypothetical treatment preferences for surgery or imiquimod for LM using standard gamble technique. | Questionnaire completed at 12 weeks post surgery (follow up visit)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Marsden, Dr, Principal Investigator — University Hospital Birmingham NHS Foundation Trust
Locations (1):
- Dr J Marsden, Queen Elizabeth Hospital, Birmingham, United Kingdom